CLINICAL TRIAL: NCT06530732
Title: Deep Cervical Lymphatlc-Venous Anastomosis Surgery for the Treatment of Alzheimer's Disease: A Pilot Study (DIVA Study)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2024106
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — lecanemab

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): receiving dcLVA surgery plus standard medication
  Interventions: Procedure: Deep Cervical lymphatlc-Venous Anastomosis Surgery; Drug: Lecanemab
- control group (Active Comparator): receiving standard medication alone
  Interventions: Drug: Lecanemab

INTERVENTIONS:
Procedure: Deep Cervical lymphatlc-Venous Anastomosis Surgery — Cervical deep lymphatic-venous anastomosis (dcLVA) can promote the flow of cerebrospinal fluid within the glymphatic system. The procedure involves connecting deep cervical lymphatic vessels to veins, reducing pressure on lymph nodes and allowing lymphatic fluid from high-pressure vessels to flow into the lower-pressure venous system. This surgical intervention enhances the clearance of waste in the glymphatic system, particularly amyloid-beta (Aβ) and tau proteins. By facilitating the removal of these AD-associated proteins from the brain, dcLVA can reduce local tissue fibrosis and cervical nerve compression, potentially reversing degenerative changes, slowing disease progression, and improving the quality of life for AD patients.
  Arms: experimental group
Drug: Lecanemab — The newly approved anti-beta-amyloid (Aβ) monoclonal antibody Lecanemab can delay AD progression but is only suitable for patients in the early stages. For those with moderate to severe AD, Lecanemab is not effective.

SUMMARY:
The goal of this clinical trial is to To demonstrate the Safety and Efficacy of dcLVA Surgery for the Treatment of Alzheimer's Disease. Patients who meet the inclusion and exclusion criteria and consent to participate will be randomly assigned to either the experimental group (receiving dcLVA surgery plus standard medication) or the control group (receiving standard medication alone)

Participants will:

Undergo cognitive assessment and brain MRI assessment; Undergo a lumbar puncture; Undergo an injection of 20ml of gadodiamide contrast agent at a concentration of 0.5 mmol/L (1ml gadodiamide: 20ml 0.9% saline).

Primary Outcome Measures: The change in the sum of Clinical Dementia Rating Scale (CDR) scores at 12-month in relative to baseline

DETAILED DESCRIPTION:
This study aims to enroll patients diagnosed with AD. Patients who meet the inclusion and exclusion criteria and consent to participate will be randomly assigned to either the experimental group (receiving dcLVA surgery plus standard medication) or the control group (receiving standard medication alone). Following randomization, patients will undergo cognitive and brain MRI assessments, a lumbar puncture, and an injection of 20ml of gadodiamide contrast agent at a concentration of 0.5 mmol/L (1ml gadodiamide: 20ml 0.9% saline). MRI imaging scans will be conducted at 4 hours, 24 hours, and 48 hours post-injection to measure the dural signal unit ratio, which will be used to assess glymphatic clearance function. The study will track changes in cognitive function and glymphatic clearance function at baseline and during follow-up periods (7 days post-surgery, 6 months, and 12 months) and will evaluate the safety of the two treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as an AD patient according to biological markers and clinical symptoms;
* Over 35 years old and with an MMSE or MOCA score ≤ 26;
* The patient or family member has signed an informed consent form.

Exclusion Criteria:

* Inability to cooperate with lumbar puncture;
* Cognitive impairment due to neurological infections (e.g., HIV, neurosyphilis, autoimmune encephalitis) or systemic diseases (e.g., diabetes, thyroid dysfunction);
* Significant organ dysfunction (heart, lung, liver, kidney);
* Coagulation disorders or contraindications to surgery;
* Inability to fully cooperate with follow-up visits.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The rate of change in the total score of the Clinical Dementia Rating Scale | Time Frame: baseline,7 days post-surgery,3-month,6-month and 12-month
  The change in the sum of Clinical Dementia Rating Scale (CDR) scores at 12-month in relative to baseline , using the Chinese version of the CDR scale, with a score range of 0-3 points for each item.The total score ranges from a minimum of 0 points to a maximum of 18 points, where a higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No